CLINICAL TRIAL: NCT05149612
Title: The Effect of Heat Therapy on Shoulder Pain and Physiologic Parameters After Laparoscopic Cholecystectomy: A Randomized Controlled Trail
Brief Title: The Effect of Heat Therapy on Shoulder Pain and Physiologic Parameters After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hanife DURGUN, PhD, RN, Assistant Professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: cholecystectomy
Record Dates: First submitted 2021-11-26; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Cholecystectomy; Nursing Caries; Shoulder Pain
Keywords: hot application; postoperative pain; nursing care; laparoscopic cholecystectomy
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative | interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: The individuals in the sample group will be divided into two groups as the hot application group and the control group. Individuals in the control group will not be treated with heat.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be told which group they are in. In order to avoid bias in the data collection phase, support will be received from the nurses working in the general surgery service independently of the research, and from the independent statistical expert, apart from the researcher, in the database of the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat Therapy Group (Experimental): The patients in the intervention group will be treated with hot water bags twice, for 20 minutes in the morning and 20 minutes in the evening, to the shoulder area, starting four hours after the operation, until the patient is discharged.
  Interventions: Other: Heat Therapy
- Control group (No Intervention): When the individuals in the control group have pain, analgesic drug treatment will be applied at the request of the physician, and no other intervention will be applied.

INTERVENTIONS:
Other: Heat Therapy — Patients in the intervention group will be treated with hot water bags twice, 20 minutes in the morning and 20 minutes in the evening, starting four hours after the operation until discharge. In accordance with the literature, the water bag filled with 55 ± 2°C hot water will be wrapped with 2 towels. The water bag will be applied to the shoulder area while the patient is in the fawler or semi-fawler position. After 20 minutes, the hot application will be terminated. Pain and physiological parameters of the patients will be evaluated at the 0th minute, 30th minute, 4th hour, 12th hour, 24th hour and 48th hour postoperatively. At the same time, when individuals have pain, analgesics will be administered at the request of the physician.
  Arms: Heat Therapy Group

SUMMARY:
This study was planned to determine the effect of hot application applied to patients undergoing laparoscopic cholecystectomy on shoulder pain and physiological parameters (blood pressure, pulse, respiratory rate, pain score, oxygen saturation.

The hypothesis of the study: To see the effect of hot application and its effect on physiological parameters after hot application in individuals who have undergone laparoscopic cholecystectomy.

The population of the study will consist of patients who were admitted to the OMU SUVAM General Surgery Service and underwent laparoscopic cholecystectomy.

The sample of the study will consist of individuals who have undergone 84 laparoscopic cholecystectomy operations, who agreed to participate in the study, and who met the criteria for inclusion in the study, between the specified dates.

The sample size of the study was determined in the G*Power 3.1.9.4 program by considering Cohen's standard effect sizes. Effect size was calculated based on 0.25, Type I error 0.05, Type II error 0.20 (80% power) and 38 patients were calculated for each group, but considering data loss, it was aimed to reach 10% more, with 42 patients for each group and 84 patients in total.

Which group the individuals in the sample group would be in was determined by randomization, and a randomization table was created over two groups.

In the study, data will be collected using the Patient Information Form, Visual Analogue Scale (VAS) and Physiological Parameter Form.

The patients in the intervention group will be treated with hot water bags twice, for 20 minutes in the morning and 20 minutes in the evening, to the shoulder area, starting four hours after the operation, until the patient is discharged.

When the individuals in the control group have pain, analgesic drug treatment will be applied at the request of the physician, and no other intervention will be applied.

DETAILED DESCRIPTION:
In the management of shoulder pain experienced by individuals after laparoscopic cholecystectomy, pharmacological methods such as nonsteroidal anti-inflammatory drugs (NSAID), gabapentinoids, local analgesics, cyclooxygenase-2 (COX-2) inhibitors, transversus abdominis plane (TAP) block and opioids (Eftekhariyazdi et al. 2020; Gurusamy et al. 2014; Salazar-Perra et al. 2020) and peripheral techniques, cognitive behavioral techniques, and non-pharmacological methods other than these can be applied in order to increase the effectiveness of pharmacological methods or to increase the effectiveness of pharmacological methods (İbrahim and Ali 2020; Komann et al. et al. 2020; Pak et al. 2016; Tick et al. 2018; Şimsek Wild 2019).

One of the techniques commonly used to reduce or relieve pain among peripheral techniques is hot application. Hot application activates the gate control mechanism, stimulates tactile receptors, removes metabolic wastes, increases the release of endorphins, reduces muscle spasms as a result of the change in viscoelastic properties in tissues, reduces pressure, tension and hypoxia in nerve endings, raises the pain threshold, provides sedation and relaxes the individual. it reduces or relieves pain (Ibrahim and Ali 2020; Perry et al. 2017). In order to benefit from the therapeutic effect of hot application, the application time should not exceed 30 minutes. If the application period lasts more than 35-40 minutes, congestion occurs in the tissue, and in hot applications lasting more than one hour, vasoconstriction may occur instead of vasodilation, and the opposite of the desired effect may occur. In hot application, the temperature is as important as the time. Although there is no evidence-based guideline for hot applications, the temperature should be 40-45ºC.

It is recommended that hot application at these temperatures has a therapeutic effect by giving heat to the skin (Ibrahim and Ali 2020; Türkmen 2017). In addition, it has an important place in nursing practices as one of the preferred nursing interventions in the non-pharmacological treatment of pain due to its ease of use, high level of patient satisfaction and rare side effects (Mohamed 2016; Perry et al. 2017).

Although there are studies in the literature in which different non-pharmacological nursing interventions have been applied to manage the shoulder pain experienced by individuals after cholecystectomy, no study has been found in which warm application has been made. Therefore, this study was planned to examine the effect of hot application applied to patients who underwent laparoscopic cholecystectomy on shoulder pain and physiological parameters.

This study was planned to determine the effect of hot application applied to patients undergoing laparoscopic cholecystectomy on shoulder pain and physiological parameters.

The hypotheses of the study:

H01: Warm application applied after laparoscopic cholecystectomy is not effective in reducing shoulder pain experienced by individuals.

H11: Warm application applied after laparoscopic cholecystectomy reduces the shoulder pain experienced by individuals.

H02: Warm application applied after laparoscopic cholecystectomy is not effective in maintaining the physiological parameters of individuals within normal limits.

H12: Warm application applied after laparoscopic cholecystectomy ensures that the physiological parameters of the patients are maintained within normal limits.

ELIGIBILITY:
Inclusion Criteria:

* who agreed to participate in the research
* 18 years old and over
* BMI within normal limits
* VAS score of 5 or higher

Exclusion Criteria:

* who refused to participate in the research
* with a history of upper laparotomy
* Having endocrine, renal, hepatic or immunological disease
* ASA (American Society of Anesthesiologists) score above 3
* with chronic shoulder pain
* Regular use of analgesics
* using sedative drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Pain Score | At the 0th minute right after the patients come from the operation
  The primary outcome of the study was to measure pain using a 10-cm VAS, with high numbers meaning greater pain intensity. The VAS is used to measure various subjective clinical phenomena, including pain. It is quick and easy to use and score. The 0-10 VAS requires the patients to choose a number from 0 to 10 that best represents their pain; 0 is the equivalent of "no pain," and 10 is the equivalent of the worst imaginable pain
Pain Score | At the 30th minute after the patients come from the operation
  The primary outcome of the study was to measure pain using a 10-cm VAS, with high numbers meaning greater pain intensity. The VAS is used to measure various subjective clinical phenomena, including pain. It is quick and easy to use and score. The 0-10 VAS requires the patients to choose a number from 0 to 10 that best represents their pain; 0 is the equivalent of "no pain," and 10 is the equivalent of the worst imaginable pain
Pain Score | At the 4th hour after the patients come from the operation,
  The primary outcome of the study was to measure pain using a 10-cm VAS, with high numbers meaning greater pain intensity. The VAS is used to measure various subjective clinical phenomena, including pain. It is quick and easy to use and score. The 0-10 VAS requires the patients to choose a number from 0 to 10 that best represents their pain; 0 is the equivalent of "no pain," and 10 is the equivalent of the worst imaginable pain
Pain Score | At the 12th hour after the patients come from the operation
  The primary outcome of the study was to measure pain using a 10-cm VAS, with high numbers meaning greater pain intensity. The VAS is used to measure various subjective clinical phenomena, including pain. It is quick and easy to use and score. The 0-10 VAS requires the patients to choose a number from 0 to 10 that best represents their pain; 0 is the equivalent of "no pain," and 10 is the equivalent of the worst imaginable pain
Pain Score | At the 24th hour after the patients come from the operation
  The primary outcome of the study was to measure pain using a 10-cm VAS, with high numbers meaning greater pain intensity. The VAS is used to measure various subjective clinical phenomena, including pain. It is quick and easy to use and score. The 0-10 VAS requires the patients to choose a number from 0 to 10 that best represents their pain; 0 is the equivalent of "no pain," and 10 is the equivalent of the worst imaginable pain
pain Score | At the 48th hour after the patients come from the operation
  The primary outcome of the study was to measure pain using a 10-cm VAS, with high numbers meaning greater pain intensity. The VAS is used to measure various subjective clinical phenomena, including pain. It is quick and easy to use and score. The 0-10 VAS requires the patients to choose a number from 0 to 10 that best represents their pain; 0 is the equivalent of "no pain," and 10 is the equivalent of the worst imaginable pain

CONTACTS AND LOCATIONS:
Overall Officials: Hanife Durgun, PhD, Principal Investigator — Ordu University
Locations (1):
- Ordu Üniversitesi, Ordu, Altınordu, Turkey (Türkiye)